CLINICAL TRIAL: NCT00294944
Title: The Effectiveness of Idazoxan in Treating TRD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SHEBA-05-3911-JZ-CTIL
Record Dates: First submitted 2006-02-19; First posted 2006-02-22 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Idazoxan

INTERVENTIONS:
Drug: Idazoxan

SUMMARY:
Assessing the effectiveness of Idazoxan as a treatment for depressive patients who did not respond to treatment with SSRI

ELIGIBILITY:
Inclusion Criteria:

* MDD patients
* Did not respond to at least one treatment of 4-6 weeks of SSRI in adequate dose
* In or out patients

Exclusion Criteria:

* Psychotic symptoms

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel